CLINICAL TRIAL: NCT01808391
Title: A Prospective Multicenter Post Approval Study to Evaluate the Long-term Safety and Efficacy of the Resolute Integrity in the Japanese All-comers Patients With Coronary Artery Disease
Brief Title: A Prospective Multicenter Post Approval Study to Evaluate the Long-term Safety and Efficacy of the Resolute Integrity in the Japanese All-comers Patients With Coronary Artery Disease (PROPEL)
Status: Completed | Type: Observational
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: PROPEL version 3.0 - AEEI
Record Dates: First submitted 2013-03-04; First posted 2013-03-11 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease; Drug-eluting Stent
Keywords: Coronary artery disease; Heart disease; Myocardial ischemia; Cardiovascular disease; Arteriosclerosis; Vascular disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clinical Follow-up Cohort: The clinical FU cohort comprises among patients who underwent clinical FU at 9, 12, and 24 months after index PCI those who arbitrarily underwent angiographic FU at 22 months (±60 days) after index PCI and those who did not undergo angiographic follow-up at all during the entire study period.
- Routine Angiographic Follow-up Cohort: The routine angiographic FU cohort comprises patients who underwent clinical FU at 9, 12, and 24 months after index PCI those who undergo angiographic FU at 10 months (±60 days) after index PCI.

SUMMARY:
This is a prospective, multicenter, historical controlled study. The present clinical study will measure non-inferiority of 12 month TLF rate compared to historical control.The selected historical control is the Xience V arm from RESOLUTE All-Comer clinical study, that study is a prospective, multicenter, randomized, two-arm, international, open-label study.The historical control did not have angiographic follow up before 12 months, in the present clinical study, only subjects with clinical follow-up conducted at 12 months without any pre-specified angiographic assessment prior to 12 month clinical follow-up will be part of this analysis cohort. Out of the total 1200 patients, 900 patients (clinical follow-up cohort) will be included in this analysis cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older.
* Patients with symptomatic coronary disease.
* Patients with a clinical indication for PCI and stenting of at least one coronary lesion, visually confirmed on coronary angiography.
* Patients who give informed consent to participate in this clinical study and sign the informed consent form approved by the institutional review board of each study site before the index PCI.
* Patients who agree to undergo all clinical follow-up procedures specified in the protocol for this clinical study.
* Patients in whom more than 50% occlusion or stenosis is visually confirmed in a native coronary artery with a diameter of 2.5 mm - 3.5 mm on coronary angiography and that has an anatomical structure suitable for PCI using Resolute Integrity zotarolimus-eluting stent.

Exclusion Criteria:

* Patients aged 85 years or older.
* Patients with cardiogenic shock.
* Patients who are pregnant or possibly pregnant.
* Patients who cannot comply with the antiplatelet therapy specified for this clinical study.
* Patients scheduled to undergo elective surgery within 6 months post-index PCI.
* Patients with a history of allergic reaction or hypersensitivity to zotarolimus, sirolimus, tacrolimus, everolimus, or other analogues or derivatives.
* Patients with an allergic reaction to antiplatelet or anticoagulant drugs, such as heparin, aspirin, ticlopidine, or clopidogrel, or contrast agents, or those who cannot tolerate these substances and to whom appropriate treatments cannot be given.
* Patients with hypersensitivity to cobalt, nickel, chrome, molybdenum, coated polymer (e.g., BioLinx) contained in the materials of the study device or in whom these substances are specifically contraindicated.
* Patients who are currently participating in a clinical study of another drug or medical device and in whom assessment of the primary endpoint of that study has not been completed or clinically interferes with the endpoints of this clinical study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Among 1,200 patients to be registered at the website database, the first 900 continuously registered patients will be then assigned to the clinical follow-up cohort, and the remaining 300 patients to the routine angiographic follow-up cohort.
Sampling Method: Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
TLF (target lesion failure) | 12 months
  The composite of Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel) or Target Lesion Revascularization (TLR; clinically indicated) (= device oriented endpoint).

SECONDARY OUTCOMES:
Delivery success | stent implantation until hospital discharge (average 1-5 days)
  Complete passage of the stent across the target lesion with full expansion of the stent to the desired diameter at the desired location.
  Note:
  Failed delivery: failure to pass the stent through the guiding catheter into the coronary artery,failure to pass it completely across the target lesion, or failure to expand the stent to its desired diameter. Failed delivery includes proximal deployment defined as those instances of failed delivery when the stent could be advanced only partially across the target lesion but was deployed nonetheless by full expansion.
Lesion success | stent implantation until hospital discharge (average 1-5 days)
  Lesion success defined as the attainment of a less than 50% residual stenosis by any percutaneous method.
TLF (target lesion failure) | 30 days, 6, 9, 12, 24 and 36 months after index PCI
  The composite of Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel) or Target Lesion Revascularization (TLR; clinically indicated) (= device oriented endpoint).
TVF (target vessel failure) | 30 days, 6, 9, 12, 24 and 36 months after index PCI
  The composite of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization by percutaneous or surgical methods.
MACE (major adverse cardiac event) | 30 days, 6, 9, 12, 24 and 36 months after index PCI
  All-cause death, myocardial infarction (QWMI and NQWMI), emergency coronary artery bypass graft(CABG), or TLR by medical or surgical procedure.
Stent thrombosis | 30 days, 6, 9, 12, 24 and 36 months after index PCI
  Incidence of ARC-defined "definite" and "probable" stent thrombosis, and the combined incidence of "definite/probable" stent thrombosis.
Duration of dual antiplatelet therapy | 12, 24 and 36 months after index PCI
  Duration of DAPT after index PCI including the reason for interruption and discontinuation.
Cerebrovascular accident | 30 days, 6, 9, 12, 24 and 36 months afetr index PCI
  1. Neurological disorder that appears rapidly and persists for at least 24 hours, and is attributable to a reduction in the cerebrovascular blood flow due to bleeding or ischemia.
  2. If an AE due to CVA occurs, it is desirable to obtain diagnostic imaging findings constituting evidence or a diagnosis by a specialist.
  3. TIA of which the symptoms disappear within 24 hours is not CVA.
Procedure success | stent implantation until hospital discharge (average 1-5 days)
  The attainment of < 50%, residual stenosis of the target lesion and no in-hospital MACE as reported by the physician.

OTHER OUTCOMES:
Comparison of long-term clinical outcomes due to a difference in follow-up procedure (clinical follow-up or routine angiographic follow-up) after index PCI. | 24 months after index PCI
Evaluation of medical economics | 24 months after index PCI
  The objectives of this clinical study are to 1) assess the efficacy and safety of RI-ZES at 10 and 22 months (±60 days) after index PCI for routine angiographic FU after index PCI and to 2) investigate its medical costs.

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, MD, Principal Investigator — Toho University Medical Center Ohashi Hospital
Locations (1):
- Non-profit organization Associations for Establishment of Evidence in Interventions, Minato-ku, Tokyo, Japan